CLINICAL TRIAL: NCT07354399
Title: Resistance Training Among Women With Coronary Artery Disease
Brief Title: Resistance Training Added to Aerobic Interval Training to Improve Aerobic Capacity and Muscle Mass in Women With Coronary Artery Disease
Acronym: VAKAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Borut Jug, Professor, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UKCLRehabVAKAR
Record Dates: First submitted 2025-12-08; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease With Myocardial Infarction
Keywords: Coronary Artery Disease; Resistance Training; Cardiac Rehabilitation; Women
MeSH Terms: conditions — Coronary Artery Disease, Autosomal Dominant, 1; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Interval Training (Active Comparator)
  Interventions: Other: Aerobic Interval Training
- Combined Training 1 (Experimental)
  Interventions: Other: Aerobic Interval Training; Other: Traditional Resistance Training
- Combined Training 2 (Experimental)
  Interventions: Other: Aerobic Interval Training; Other: Prolonged Eccentric Phase Resistance Training

INTERVENTIONS:
Other: Aerobic Interval Training — Interval cycling, performed at 70-80% of the heart rate reserve (HRR) as determined during the cardiopulmonary exercise test. The training is structured as alternating high- and low-intensity intervals.
Other: Traditional Resistance Training — Resistance training with traditional tempo (1-second ascent, 2-second descent) - squat exercise and horizontal pull.
  Arms: Combined Training 1
Other: Prolonged Eccentric Phase Resistance Training — Resistance training with prolonged eccentric phase tempo (1-second ascent, 5-second descent) - squat exercise and horizontal pull.
  Arms: Combined Training 2

SUMMARY:
The goal of this clinical trial is to find out whether partly replacing aerobic interval training (AIT) with resistance training (RT) leads to greater improvements in physical fitness and muscle mass in women with coronary artery disease (CAD) during cardiac rehabilitation.

The main questions this study aims to answer are:

* Does combining RT (squats and pulling exercises with weights) with a reduced amount of AIT (cycling) improve aerobic fitness in the same way as AIT alone?
* Does the combined training lead to greater improvements in muscle mass compared with AIT alone?
* Does slow-speed RT (slower lowering phase) result in lower heart rate and blood pressure during exercise compared with normal-speed RT?

Researchers will compare three exercise programs:

* AIT only (control group),
* AIT combined with normal-speed RT (1-second lifting, 2-second lowering),
* AIT combined with slow-speed RT (1-second lifting, 5-second lowering).

Participants will take part in a 12-week cardiac rehabilitation program and will train three times per week.

At the start and end of the program, participants will complete a cycling fitness test, body composition assessment, blood sampling, two strength tests, and quality-of-life questionnaire.

DETAILED DESCRIPTION:
CAD remains one of the leading causes of death among women worldwide. Although cardiac rehabilitation programs with AIT are well established, the optimal way to include RT in this population remains unclear. Historically, RT was limited in patients with heart disease due to concerns about excessive blood pressure responses and cardiovascular risk. However, recent evidence shows that properly prescribed RT is safe and may significantly improves muscle strength, aerobic fiitness, and overall quality of life.

The study consists of two sequential phases. The first is a crossover feasibility phase designed to compare the acute hemodynamic responses (blood pressure, heart rate) and rate of perceived exertion between two RT protocols: (1) traditional high-load RT (1-second lift, 2-second descent) and (2) high-load RT with a prolonged eccentric phase (1-second lift, 5-second descent). The goal of this phase is to confirm the feasibility and short-term safety of both approaches before inclusion in the main trial.

The second phase is a three-arm, parallel-group randomized controlled trial. After baseline assessments, participants are randomized into one of three groups using block randomization with variable block sizes to ensure balanced allocation throughout recruitment.

The 12-week intervention includes three supervised sessions per week, totaling 36 visits. AIT follows a structured progression based on heart rate reserve, alternating between high- and low-intensity cycling intervals on a stationary ergometer. RT sessions consist of compound lower-body and upper-body movements (hex-bar squat and horizontal cable pull), performed at approximately 80% of one-repetition maximum. Training intensity, load progression, and repetition tempo are standardized across groups, ensuring equivalent time under tension per set.

To maintain participant safety, all exercise sessions are supervised by medical and rehabilitation staff, including a physiotherapist, nurse, and kinesiologist, with a cardiologist on call. Continuous heart rate monitoring and pre- and post-exercise blood pressure measurements are performed during each session. Any adverse events will be recorded and reviewed by the study physician.

Statistical analyses will follow the intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* documented CAD,
* stable clinical status (at least 1 month since myocardial infarction and/or elective percutaneous coronary intervention, at least 3 months since cardiac surgery).

Exclusion Criteria:

* based on the American Heart Association guidelines for resistance training in patients with CAD,
* pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Maximal Aerobic Capacity | From enrollment to the end of treatment at 12 week.
  Maximal aerobic capacity (VO2peak) will be assessed using a modified Ramp protocol on the Schiller ERR 911 cycle ergometer in combination with the Cardiovit CS-200 Excellence ergo-spirometer (Schiller, Switzerland). Following baseline spirometry, participants will perform a warm-up phase of unloaded cycling for up to three minutes, after which the workload will increase incrementally by 10-25 W every minute until exhaustion or the appearance of clinical indications for test termination. Throughout the test, the supervisor will monitor for any signs or symptoms warranting termination, in accordance with the American Heart Association guidelines.
Lean Body Mass | From enrollment to the end of treatment at 12 weeks.
  Body composition, including lean body mass (also called fat-free mass; calculated by subtracting body fat weight from total body weight) and fat mass, will be assessed using whole-body dual-energy X-ray absorptiometry (DXA) (Hologic, USA), which is considered the gold standard for evaluating body composition due to its high accuracy and reproducibility .

SECONDARY OUTCOMES:
Blood Biomarkers | From enrollment to the end of treatment at 12 weeks.
  As part of routine clinical blood draws, fasting blood samples will be obtained before the first and last training sessions. They will be analysed for standard clinical parameters (including blood lipids and others).
Handgrip Strength | From enrollment to the end of treatment at 12 weeks.
  Handgrip strength will be assessed using a hand dynamometer (Jamar). Participants will hold the dynamometer with the arm alongside the body and the elbow flexed at 90 degrees, and will be instructed to squeeze as hard as possible for 3-5 seconds. Three measurements will be performed for each hand, with 1 minute of rest between trials. The highest value obtained will be used for analysis.
30-Second Sit-to-Stand Test | From enrollment to the end of treatment at 12 weeks.
  Lower-limb functional strength will be assessed using the 30-second sit-to-stand test. Participants rise from and return to a seated position as many times as possible within 30 seconds, using a standard chair (43 cm) without armrests, with arms crossed over the chest and feet flat on the floor. The outcome is the number of fully completed stands in 30 seconds. If the participant is unable to stand without using the arms, the score is recorded as 0.
Quality of Life Measure | From enrollment to the end of treatment at 12 weeks.
  Health-related quality of life will be assessed using the Heart Quality of Life Questionnaire (HeartQoL). The questionnaire yields scores ranging from 0 to 3, with higher scores indicating better health-related quality of life. The overall HeartQoL score is calculated as the mean of all item responses and includes one global scale and two subscales (physical and emotional).

CONTACTS AND LOCATIONS:
Overall Officials: Borut Jug, MD, Ph.D., Principal Investigator — University Medical Centre Ljubljana, Slovenia
Locations (1):
- University Medical Centre Ljubljana (Department of Vascular Diseases, Division of Internal Medicine), Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hansen D, Abreu A, Doherty P, Voller H. Dynamic strength training intensity in cardiovascular rehabilitation: is it time to reconsider clinical practice? A systematic review. Eur J Prev Cardiol. 2019 Sep;26(14):1483-1492. doi: 10.1177/2047487319847003. Epub 2019 May 2. PMID 31046441
- [Background] Terada T, Pap R, Thomas A, Wei R, Noda T, Visintini S, Reed JL. Effects of muscle strength training combined with aerobic training versus aerobic training alone on cardiovascular disease risk indicators in patients with coronary artery disease: a systematic review and meta-analysis of randomised clinical trials. Br J Sports Med. 2024 Oct 22;58(20):1225-1234. doi: 10.1136/bjsports-2024-108530. PMID 39214675
- [Background] Kambic T, Sarabon N, Hadzic V, Lainscak M. Effects of high- and low-load resistance training in patients with coronary artery disease: a randomized controlled clinical trial. Eur J Prev Cardiol. 2022 Nov 8;29(15):e338-e342. doi: 10.1093/eurjpc/zwac063. No abstract available. PMID 35512240
- [Background] Douglas J, Pearson S, Ross A, McGuigan M. Chronic Adaptations to Eccentric Training: A Systematic Review. Sports Med. 2017 May;47(5):917-941. doi: 10.1007/s40279-016-0628-4. PMID 27647157